CLINICAL TRIAL: NCT06617663
Title: Online Therapy Youth, Equivalent to Treatment As Usual?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GGZ Noord-Holland-Noord (Other)
Collaborators: UMC Utrecht (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GGZNHNETB2024
Record Dates: First submitted 2024-05-27; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-08

CONDITIONS: Depression; Trauma; Compulsive Disorder; Anxiety; Unexplained Symptom, Medically
Keywords: EMDR intervention; ACT internvention; youth 12.18
MeSH Terms: conditions — Depression; Wounds and Injuries; Compulsive Personality Disorder; Anxiety Disorders; Medically Unexplained Symptoms | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Intervention Model Description: A randomized non-inferiority design will be used to demonstrate whether or not online treatment is inferior to treatment as usual (TAU). Data will be analyzed according to the intention-to-treat principle, with all randomized clients included in the analysis, as well as "per protocol" (where a minimum of 12 sessions must be completed).
  In both the intention-to-treat and "per protocol" analyses, mixed general linear (or nonlinear, depending on score distribution) models will be performed, where the main effect of treatment and the interaction between effect and treatment setting are our main measures of interest. Mixed models have the advantage that they 1) account for multiple measures within the same individual, and 2) account for missing values. All analyses are adjusted for baseline value on the outcome measure, gender, and age. To detect age- and gender-specific effects, analyses will also be performed separately by gender and age group.
Who Masked: Participant, Care Provider
Masking Description: Block randomization will be conducted by an independent researcher who is not involved in the study assessments or therapies. This process will assign clients to either online or in-patient treatment to ensure approximately equal distributions of individuals aged 12-15 and 15-18, as well as balanced representation of different sexes. For both video call treatment and treatment at a physical location, the waiting time until the start of treatment will be the same; treatment will begin within a maximum of 2 months from registration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- EMDR online (Experimental): The investigators will use the Association for EMDR (called VEN in the Netherlands) protocol for individuals up to age 18 through videoconferencing with a therapist, supported by MOOVD as a digital intervention platform.
  Interventions: Behavioral: EMDR
- EMDR on-site (Active Comparator): The investigators will use the Association for EMDR (called VEN in the Netherlands) protocol for individuals up to age 18 at a physical location . Various working memory load techniques may be used, including the light bar.
  Interventions: Behavioral: EMDR
- ACT online (Experimental): ACT, along with an e-health program, will be offered through video conferencing.
  Interventions: Behavioral: ACT
- ACT on-site (Active Comparator): ACT will be offered at a physical location without additional e-health modules.
  Interventions: Behavioral: ACT

INTERVENTIONS:
Behavioral: EMDR — Eye Movement Desensitization and Reprocessing (EMDR) is a therapy designed to alleviate the distress associated with traumatic memories.
  Arms: EMDR on-site; EMDR online
Behavioral: ACT — Acceptance and Commitment Therapy (ACT) is an action-oriented approach to psychotherapy that stems from traditional behavior therapy and cognitive behavioral therapy. Clients learn to stop avoiding, denying, and struggling with their inner emotions and, instead, accept that these deeper feelings are appropriate responses to certain situations and should not prevent them from moving forward in their lives. The ACT Your Way method is specifically designed for young people.
  Arms: ACT on-site; ACT online

SUMMARY:
With growing waiting lists in specialized youth mental health care (sGGZ) and shortages of care staff, finding creative solutions to respond to this scarcity issue is important. Online treatment is an example of this, which, especially for young people growing up in a digital age, can be an appropriate and accessible alternative to treatment at a physical location. Online treatment via video calling among youth, while researched and proven effective in a blended form, has not yet been sufficiently researched as a complete replacement for treatment at a physical location. As a result, the potential added value of online treatment for the pressing scarcity issue in healthcare is not yet sufficiently clear.

This study therefore focuses on investigating the effectiveness of fully online treatment using two proven effective interventions: Eye Movement Desensitization and Reprocessing (EMDR) and Acceptance and Commitment Therapy (ACT) within the youth sGGZ. With the results of this research at GGZ-NHN, the investigators want to contribute to the development of guidelines and standards for the implementation of online treatments within Dutch youth mental health care.

DETAILED DESCRIPTION:
In recent years, there has been tension between young people's need for specialty mental health care (sGGZ) and the lack of sufficient available resources and staff. As a result, waiting lists have increased. To increase the accessibility and efficiency of care, online treatment through video calling is a promising method. Online treatment can help reduce waiting lists, as there are no limitations in terms of physical space and geographical proximity to clients and health care professionals, and it allows mental health professionals to work more efficiently and reach more young people, as they have no travel time and can plan flexibly from any location. An additional advantage of online treatment is its low threshold. Young people with mental health problems often face stigma and shame for physically going to a mental health facility. Online treatment via video call can remove this barrier and allow young people to access the care they need from their familiar surroundings.

It is plausible that fully online treatment with youth is at least as effective as treatment in a physical location, regardless of cultural origin, gender, or social environment, because youth are familiar with digital communication, the technical application has now been sufficiently developed, and blended treatment has been assessed as effective in research. However, it has not yet been sufficiently scientifically studied whether fully online treatment via video calling in youth is actually a worthy alternative to physical treatment in reducing mental health problems among youth.

This research project of GGZ Noord-Holland-Noord (GGZ-NHN), on which Drs. E. te Brake will receive her doctorate, therefore focuses on the effectiveness of fully online treatment within the youth sGGZ compared to regular treatment at a physical location. This study explicitly includes a role for experts by experience who, from the perspective of clients and relatives, contribute to the design and execution of the study and the implementation of the results into treatment practice.

The proposed research includes a Randomized Controlled Trial (RCT), specifically focused on two common therapies with adolescents in the sGGZ: Acceptance and Commitment Therapy (ACT) and Eye Movement Desensitization and Reprocessing (EMDR). Cognitive behavior therapy (CBT) could be an obvious choice because of its extensive knowledge and experience, as well as available scientific evidence. But the investigators prefer the more generalist ACT because CBT uses a separate protocol for each target group. As a third-generation form of therapy, ACT is a suitable intervention because its universal protocol is applicable to a broad target group. Moreover, ACT has been shown to be not inferior to cognitive behavioral therapy in terms of effectiveness. The methodology shows significant improvements in depressive symptoms, quality of life, and perception of competence.

Treatment will be protocolized according to the guidelines prescribed by the manual for this purpose. The protocol used is specifically intended for the target group aged 15-25. However, it is known that adolescents between 12 and 15 can also benefit well from ACT. Age-appropriate adjustments in language use will be applied here. In addition, EMDR will be investigated for trauma-specific symptoms, as digital tools are available with EMDR that allow for a good comparison with EMDR in a physical location.

Because an RCT generates reliable and generalizable information, and the investigators examine two commonly used interventions in the mental health system, the study fits well with policymakers' effectiveness-evidence criteria. If it turns out that fully online treatment is a worthy alternative to treatment at a physical location, then this lays a foundation for online work. It thus contributes to the low threshold, accessibility, and affordability of youth mental health care.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 12-18 years who would benefit from ACT or EMDR within the SGGZ, as determined by the screeners at registration or current primary practitioner.
* Client is stable, i.e. there is no serious crisis (to be determined by screener cq primary practitioner)
* Sufficient command of the Dutch language to complete the questionnaires.
* Client does not participate in other (intervention) studies

Exclusion Criteria:

* Clients who are crisis-prone or enter in crisis
* Clients who are in forced care (wvggz)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Male, female
Enrollment: 172 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in the level of psychological flexibility (for the ACT arms), as measured by the AFQ-Y. | At baseline, +/- 3-months after start treatment, and at 6-months after completion of intervention (equals +/- 9 months after baseline assessment)
  Differences in psychological flexibility between individuals that receive ACT online and on-site will be measured wit the AFQ-Y. The scale has a minimum score of 0 and a maximum score of 68. A higher score indicates a greater psychological inflexibility.
Change in the degree of overall symptomatic distress, as measured by the Youth Outcome questionnaire (YOQ) | At baseline, +/- 3-months after start treatment, and at 6-months after completion of intervention (equals +/- 9 months after baseline assessment)
  Differences in symptomatic distress between treatments performed on site and those performed online will be measured with the YOQ. The questionnaire has a minimum score of 0 and a maximum score of 120. A higher scores indicate a greater level of distress.
Change in post-traumatic symptoms (for the EMDR arms), as measured by the KJTS EMDR questionnaire | At baseline, +/- 3-months within treatment, and at 6-months after completion of intervention (equals +/- 9 months after baseline assessment)
  Differences in posttraumatic stress symptoms between individuals that receive EMDR treatment on site and online will be measured with the KJTS EMDR. KJTS has a minimum score of 0 and a maximum score of 60. A higher score indicates more symptoms.
Change in the degree of societal recovery, as measured by the kidsscreen-27. | At baseline, +/- 3-months after start treatment, and at 6-months after completion of intervention (equals +/- 9 months after baseline assessment)
  It will be measured whether there is a significant difference in societal functioning between individuals who receive treatment on site and online. Minimum score is 27, maximum score is 135. Higher score indicates better societal functioning

SECONDARY OUTCOMES:
Differences in the therapeutic relationship, as measured by the WAV-12 (work alliance questionnaire) | At +/- 1 1/2 month after start treatment
  The WAV-12 will be used to examine whether there is a significant difference in therapeutic alliance between treatments performed on site and online. The minimum score of the WAV-12 , the maximum score is 60. A high score reflects a better therapeutic bond

CONTACTS AND LOCATIONS:
Locations (1):
- GGZ NHN, Alkmaar, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Midgley N, Guerrero-Tates B, Mortimer R, Edbrooke-Childs J, Mechler J, Lindqvist K, Hajkowski S, Leibovich L, Martin P, Andersson G, Vlaescu G, Lilliengren P, Kitson A, Butler-Wheelhouse P, Philips B. The Depression: Online Therapy Study (D:OTS)-A Pilot Study of an Internet-Based Psychodynamic Treatment for Adolescents with Low Mood in the UK, in the Context of the COVID-19 Pandemic. Int J Environ Res Public Health. 2021 Dec 9;18(24):12993. doi: 10.3390/ijerph182412993. PMID 34948601
- [Background] Ravens-Sieberer U, Auquier P, Erhart M, Gosch A, Rajmil L, Bruil J, Power M, Duer W, Cloetta B, Czemy L, Mazur J, Czimbalmos A, Tountas Y, Hagquist C, Kilroe J; European KIDSCREEN Group. The KIDSCREEN-27 quality of life measure for children and adolescents: psychometric results from a cross-cultural survey in 13 European countries. Qual Life Res. 2007 Oct;16(8):1347-56. doi: 10.1007/s11136-007-9240-2. Epub 2007 Aug 1. PMID 17668292
- [Background] Porter CM, Galloghly E, Burbach FR. The effective delivery of digital CBT: a service evaluation exploring the outcomes of young people who completed video conferencing therapy in 2020. The Cognitive Behaviour Therapist. 2022;15:e27. doi:10.1017/S1754470X22000216
- [Background] Pelzer, A. et al (2022), K. De balans is zoek in Jeugdzorgland. Kind Adolesc Prakt 21, 34-36
- [Background] Schueller SM, Stiles-Shields C, Yarosh L. Online Treatment and Virtual Therapists in Child and Adolescent Psychiatry. Child Adolesc Psychiatr Clin N Am. 2017 Jan;26(1):1-12. doi: 10.1016/j.chc.2016.07.011. Epub 2016 Oct 15. PMID 27837935
- [Background] Stinckens, Nele & Ulburghs, A. & Claes, Laurence. (2009). De werkalliantie als sleutelelement in het therapiegebeuren: Meting met behulp van de WAV-12, de Nederlandstalige verkorte versie van de Working Alliance Inventory. Tijdschrift Klinische Psychologie. 39. 44-60.
- [Background] Schraven, J., et al. (2023) ACT your way, kwaliteit van het protocol en eerste bevindingen van een pilot- effectonderzoek bij adolescenten met een recidiverende depressie
- [Background] caleidoZorg & CZ (2023) Tijd effectiviteit van WeMind vs. Lightbar bij EMDR-therapie in een klinische populatie
- [Background] Swain, J. et al (2015). Acceptance and Commitment Therapy for children: A systematic review of intervention studies.
- [Derived] Brake ET, Scheepers F, Mous T, Visser I, Vernhout S, Velthorst E. Comparing the effectiveness of online therapy versus in-person therapy in youth: protocol for a non-inferiority randomized controlled trial. Trials. 2025 Dec 1;27(1):3. doi: 10.1186/s13063-025-09312-9. PMID 41327248